CLINICAL TRIAL: NCT06105099
Title: One Size Does Not Fit All: From a Common Approach Towards Performance-specific Speech Intervention and Long-term Learning in Children With a Cleft Palate
Brief Title: Effect of Performance-specific Cleft Speech Intervention and Long-term Learning in Children With a Cleft Palate
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Ghent (Other)
Collaborators: Research Foundation Flanders (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 12ZO323N
Record Dates: First submitted 2023-10-02; First posted 2023-10-27 (Actual); Last update posted 2023-10-27 (Actual); Status verified 2023-10

CONDITIONS: Cleft Palate Children; Speech Disorders in Children; Cleft Lip and Palate; Speech Therapy
Keywords: Randomized controlled trial; Speech therapy; Cleft lip and palate
MeSH Terms: conditions — Cleft Lip; Communication Disorders

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Children with anterior oral cleft speech characteristics (Active Comparator): To investigate the best speech therapy approach for children with anterior oral cleft speech characteristics, we will provide three different interventions.
  Interventions: Behavioral: Motor-phonetic intervention; Behavioral: Phonological intervention; Behavioral: Combined phonetic-phonological intervention
- Children with posterior oral cleft speech characteristics (Experimental): To investigate the best speech therapy approach for children with potserior oral cleft speech characteristics, we will provide three different interventions.
  Interventions: Behavioral: Motor-phonetic intervention; Behavioral: Phonological intervention; Behavioral: Combined phonetic-phonological intervention
- Children with non-oral cleft speech characteristics (Experimental): To investigate the best speech therapy approach for children with non-oral cleft speech characteristics, we will provide three different interventions.
  Interventions: Behavioral: Motor-phonetic intervention; Behavioral: Phonological intervention; Behavioral: Combined phonetic-phonological intervention

INTERVENTIONS:
Behavioral: Motor-phonetic intervention — Children will receive phonetic articulation therapy treating consonants in a phoneme-by-phoneme basis, emphasizing phonetic placement and shaping techniques.
  Phonetic articulation therapy includes a progression of the target consonant from isolated level, syllable level, word level, sentence level, spontaneous speech level in five different steps:
  identification of the target consonant using visual, tactile, and auditory feedback techniques, discrimination between the used and targeted consonant, (3) variation and correction, (4) stabilize the target, and (5) maintenance of the target. A next level will be introduced when the child is able to correctly produce the sound in 90% of the time with minimal cues from the therapist.
Behavioral: Phonological intervention — The phonological approach consists of two phases. In the first phase, the child's attention is drawn to the contrastive features of the speech sound system which are relevant to the target consonants. Terms that describe the sound features will be introduced using words on the child's level, e.g. in the case of active nasal fricatives the words 'nose' and 'mouth' will be used. Child-friendly games will be played to illustrate the contrast between the concepts followed by activities that focus on the contrasts in non-speech sounds, in which child and therapist will alternate between being listener and speaker. At the end of this phase, minimal word pairs (e.g. tap/cap), only produced by the therapist, will be used to facilitate the child's awareness of sounds in words and meaningful differences based on distinctive features.
  In the second phase, the child will produce minimal pairs providing the opportunity to monitor his/her speech and to make self-corrections.
Behavioral: Combined phonetic-phonological intervention — Children will receive motor-phonetic articulation therapy supplemented with phonological principles. Therapy will be provided following the same five steps as the 'motor-phonetic group'. However, articulation errors will not be treated in a phoneme-by-phoneme basis. In contrast, multiple errors will be targeted simultaneously by focusing on a process. For example, if the child produces glottal stops for the /t/ and the /p/, these sounds will be treated simultaneously as sounds requiring oral front placements. Exercises will be embedded in meaningful language contexts such as minimal pairs

SUMMARY:
Speech therapy in children with a palate deals with two scientific challenges that will be addressed in this project.

The first challenge is selecting the best speech approach for a child with a specific cleft speech characteristic (CSC). Many speech therapists use a 'one-size-fits-all' approach to treat compensatory CSCs resulting in poor short- and long-term speech outcomes. To increase the effectiveness and quality of cleft speech care, it is necessary to find the best match between a specific therapy and a given type of CSC. Therefore, this proposal will compare the effect of 3 different speech approaches on the speech and quality of life in Dutch speaking children with different types of CSCs.

The second challenge is selecting the best speech approach to enhance long-term learning and transfer of newly established speech skills to untrained consonants. To date, research mainly focused on immediate therapy effects. It is unknown if permanent speech changes occur. Hence, this project will also investigate the short-term and long-term learning effects (retention and transfer) of the different speech approaches from the first objective.

This proposal will improve evidence-based and patient-tailored cleft speech therapy.

DETAILED DESCRIPTION:
Objective 1: To compare the (immediate) effect of three speech therapy approaches (i.e.

a motor-phonetic approach, a phonological approach, and a combined phonetic-phonological approach) on the speech and health-related quality of life (HRQoL) in Belgian Dutch-speaking children with a CP±L and different subtypes of compensatory CSCs (anterior oral CSCs, posterior oral CSCs, or non-oral CSCs) measured by perceptual and psychosocial outcome measures.

Objective 2: To measure the short-term effects (performance to learning) and the long-term learning effects (retention and transfer) of the three different speech therapy approaches (i.e. a motor-phonetic approach, a phonological approach, and a combined phonetic-phonological approach) on the speech and HRQoL in Belgian Dutch-speaking children with a CP±L and different subtypes of compensatory CSCs measured by perceptual and psychosocial outcome measures.

ELIGIBILITY:
Inclusion Criteria:

* Belgian Dutch-speaking children with a cleft palate with or without a cleft lip
* Aged between 4 and 12 years
* Presence of at least one compensatory speech error in their speech based on the perceptual assessment of one experienced speech-language pathologist

Exclusion Criteria:

* Children with syndromic clefts
* Oronasal fistula
* Velopharyngeal insufficiency
* Hearing disabilities based on pure tone audiometry (>25 dB HL)
* Cognitive and/or related learning disabilities or neuromuscular disorders

Ages: 4 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 135 (Estimated)
Dates: Start 2022-10-01 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Consonant proficiency | Assessment immediately pre-intervention
  Consonant proficiency will be measured in terms of percentage correctly produced consonants (%)
Consonant proficiency | Assessment immediately post-intervention
  Consonant proficiency will be measured in terms of percentage correctly produced consonants (%)
Consonant proficiency | Assessment at 1 month post-intervention
  Consonant proficiency will be measured in terms of percentage correctly produced consonants (%)
Consonant proficiency | Assessment at 3 months post-intervention
  Consonant proficiency will be measured in terms of percentage correctly produced consonants (%)
Consonant proficiency | Assessment at 6 months post-intervention
  Consonant proficiency will be measured in terms of percentage correctly produced consonants (%)

SECONDARY OUTCOMES:
Intelligibility in Context | Assessment immediately pre-intervention
  To assess possible transfer of learned speech skills to contexts outside the therapy setting, the Intelligibility in Context Scale (ICS) will be administered before and after intervention. The ICS rates the degree to which children's speech is understood by different partners (caregivers, immediate and extended family, friends, acquaintances, teachers, and strangers) on a 5-point scale (1 - never intelligible to 5 - always intelligible)
Intelligibility in Context | Assessment immediately post-intervention
  To assess possible transfer of learned speech skills to contexts outside the therapy setting, the Intelligibility in Context Scale (ICS) will be administered before and after intervention. The ICS rates the degree to which children's speech is understood by different partners (caregivers, immediate and extended family, friends, acquaintances, teachers, and strangers) on a 5-point scale (1 - never intelligible to 5 - always intelligible)
Intelligibility in Context | Assessment at 1 month post-intervention
  To assess possible transfer of learned speech skills to contexts outside the therapy setting, the Intelligibility in Context Scale (ICS) will be administered before and after intervention. The ICS rates the degree to which children's speech is understood by different partners (caregivers, immediate and extended family, friends, acquaintances, teachers, and strangers) on a 5-point scale (1 - never intelligible to 5 - always intelligible)
Intelligibility in Context | Assessment at 3 months post-intervention
  To assess possible transfer of learned speech skills to contexts outside the therapy setting, the Intelligibility in Context Scale (ICS) will be administered before and after intervention. The ICS rates the degree to which children's speech is understood by different partners (caregivers, immediate and extended family, friends, acquaintances, teachers, and strangers) on a 5-point scale (1 - never intelligible to 5 - always intelligible)
Intelligibility in Context | Assessment at 6 months post-intervention
  To assess possible transfer of learned speech skills to contexts outside the therapy setting, the Intelligibility in Context Scale (ICS) will be administered before and after intervention. The ICS rates the degree to which children's speech is understood by different partners (caregivers, immediate and extended family, friends, acquaintances, teachers, and strangers) on a 5-point scale (1 - never intelligible to 5 - always intelligible)
Health-related quality of life | Assessment immediately pre-intervention
  To evaluate the psychosocial impact of the interventions, the Velopharyngeal insufficiency Effects on Life outcomes (VELO) questionnaire will be administered before and after the intervention. This tool consists of a caregiver and child report (for children older than 8 years) addressing different domains: speech limitation, swallowing problems, situational difficulty, emotional impact, perception by others, and caregiver impact.
  The higher the score, the better the quality of life. The VELO-scores range from 0 (minimal quality of life) to 100 (maximal quality of life).
Health-related quality of life | Assessment immediately post-intervention
  To evaluate the psychosocial impact of the interventions, the Velopharyngeal insufficiency Effects on Life outcomes (VELO) questionnaire will be administered before and after the intervention. This tool consists of a caregiver and child report (for children older than 8 years) addressing different domains: speech limitation, swallowing problems, situational difficulty, emotional impact, perception by others, and caregiver impact.
  The higher the score, the better the quality of life. The VELO-scores range from 0 (minimal quality of life) to 100 (maximal quality of life).
Health-related quality of life | Assessment at 1 month post-intervention
  To evaluate the psychosocial impact of the interventions, the Velopharyngeal insufficiency Effects on Life outcomes (VELO) questionnaire will be administered before and after the intervention. This tool consists of a caregiver and child report (for children older than 8 years) addressing different domains: speech limitation, swallowing problems, situational difficulty, emotional impact, perception by others, and caregiver impact.
  The higher the score, the better the quality of life. The VELO-scores range from 0 (minimal quality of life) to 100 (maximal quality of life).
Health-related quality of life | Assessment at 3 months post-intervention
  To evaluate the psychosocial impact of the interventions, the Velopharyngeal insufficiency Effects on Life outcomes (VELO) questionnaire will be administered before and after the intervention. This tool consists of a caregiver and child report (for children older than 8 years) addressing different domains: speech limitation, swallowing problems, situational difficulty, emotional impact, perception by others, and caregiver impact.
  The higher the score, the better the quality of life. The VELO-scores range from 0 (minimal quality of life) to 100 (maximal quality of life).
Health-related quality of life | Assessment at 6 months post-intervention
  To evaluate the psychosocial impact of the interventions, the Velopharyngeal insufficiency Effects on Life outcomes (VELO) questionnaire will be administered before and after the intervention. This tool consists of a caregiver and child report (for children older than 8 years) addressing different domains: speech limitation, swallowing problems, situational difficulty, emotional impact, perception by others, and caregiver impact.
  The higher the score, the better the quality of life. The VELO-scores range from 0 (minimal quality of life) to 100 (maximal quality of life).

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Rehabilitation Sciences, Ghent, Belgium

IPD SHARING:
Plan to Share IPD: Undecided